CLINICAL TRIAL: NCT01442506
Title: Acetic Acid Guided Biopsies Compared With High Definition Endoscopy
Brief Title: Acetic Acid Guided Biopsies Compared With High Definition Endoscopy in the Detection of Barrett's Esophagus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Hoffman Arthur, principal investigator, Johannes Gutenberg University Mainz
Other Study IDs: 837.237.09
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Barrett's Esophagus
Keywords: acetic acid; virtual chromoendosopy
MeSH Terms: conditions — Barrett Esophagus | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barrett
  Interventions: Other: biopsies; Other: biopsy

INTERVENTIONS:
Other: biopsies — taking biopsies
Other: biopsy — biopsy

SUMMARY:
Specialized columnar epithelium (SCE) is considered as pathognomonic for Barrett's esophagus. Chromoendoscopy after local acetic acid application enables recognition of the mucosal surface architecture. The new available EPKi processor (Pentax, Japan) enables HD+ resolution above HDTV standard. Aim of the study is to test the efficacy of HD+ endoscopy in conjunction with i-Scan or acetic acid to diagnose Barrett's esophagus. The primary endpoint of the current prospective study is to investigate the diagnostic yield of virtual chromoendoscopy using the i scan function as compared to acetic acid chromoendoscopy and 4-quadrant biopsies.

Patients with visible columnar lined lower esophagus (CLE) are included. After standardized PPI therapy (14 days; standard dosage) patients were randomized at a 1:1 ratio to undergo either chromoendoscopy in conjunction with acetic acid application or i-Scan. Biopsies are taken in a targeted fashion using acetic acid or i scan and afterwards 4-quadrant biopsies are taken.

DETAILED DESCRIPTION:
Specialized columnar epithelium (SCE) is considered as pathognomonic for Barrett's esophagus and can be recognized by new endoscopic techniques. Aim of the study is to test the efficacy of HD+ endoscopy in conjunction with i-scan (newly developed post processing digital filter) or chromoendoscopy (acetic acid) to diagnose Barrett's esophagus.

Patients with visible columnar lined lower esophagus (CLE) or known Barrett's esophagus are included. After standardized PPI therapy (14 days; standard dosage) patients are randomized at a 1:1 ratio to undergo either chromoendoscopy in conjunction with acetic acid application (10-15ml; 1.5%) or HD+ endoscopy in conjunction with i-scan. Mucosal surface structure within CLE is graduated according to Guelrud's classification (type 1-2: endoscopic prediction: gastric epithelium; type 3-4: Barrett's epithelium). Biopsies are taken in a targeted fashion (type 1-4) in both groups and subsequently 4-quadrant biopsies were taken. Primary outcome analysis's to investigate the diagnostic yield of the different biopsy protocols.

ELIGIBILITY:
Inclusion Criteria:

* patients with CLE
* patients with known Barrett's esophagus

Exclusion Criteria:

* pregnancy
* severe coagulopathy
* known malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with suspected barrettes esophagus
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic yield of targeted biopsies with high definition endoscopy using i scan virtual chromoendoscopy and acetic acid guided biopsies | one year

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Hoffman, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- University of Mainz, Mainz, Germany

REFERENCES:
- [Derived] Hoffman A, Korczynski O, Tresch A, Hansen T, Rahman F, Goetz M, Murthy S, Galle PR, Kiesslich R. Acetic acid compared with i-scan imaging for detecting Barrett's esophagus: a randomized, comparative trial. Gastrointest Endosc. 2014 Jan;79(1):46-54. doi: 10.1016/j.gie.2013.07.013. Epub 2013 Aug 14. PMID 23953402